CLINICAL TRIAL: NCT04889664
Title: Adding Trauma-focused Psychotherapy to Ketamine Treatment for Chronic PTSD: A Pilot Study
Brief Title: Adding Trauma-focused Psychotherapy to Ketamine Treatment for Chronic PTSD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Adriana Feder, Asociate Professor Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-00167
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: PTSD
Keywords: ketamine; Written Exposure Therapy; PTSD; intervention; treatment; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine and Written Exposure Therapy (Experimental): Intravenous Ketamine 0.5 mg/kg and Written Exposure Therapy
  Interventions: Drug: Ketamine; Behavioral: Written Exposure Therapy

INTERVENTIONS:
Drug: Ketamine — Repeated intravenous Ketamine infusions.
Behavioral: Written Exposure Therapy — WET is a brief, 5-session evidence-based written trauma-focused therapy
  Other Names: WET

SUMMARY:
The current pilot project will evaluate the efficacy of adding Written Exposure Therapy (WET) to a course of repeated IV ketamine infusions in improving PTSD symptoms and maintaining symptom improvement in patients with chronic PTSD. WET is a brief, 5-session evidence-based written trauma-focused therapy without in between-session assignments, with demonstrated efficacy and low dropout rates in patients with PTSD. WET will be administered to all eligible participants; the first WET sessions will be interleaved with the last two ketamine infusions to take advantage of a window of increased neuroplasticity potentially induced by repeated ketamine infusions. WET will be administered on different days as the ketamine infusions.

DETAILED DESCRIPTION:
Current treatments for PTSD do not work for a significant proportion of individuals with PTSD, or work only partially, leaving persistent and disabling residual symptoms. The research team has led the development of ketamine for the treatment of chronic PTSD. After the initial, proof-of-concept randomized controlled trial (RCT) of a single ketamine infusion in individuals with chronic PTSD showed promising results, the study team recently completed the first RCT of repeated intravenous ketamine infusions where individuals with chronic PTSD received a course of six ketamine infusions (vs. active placebo midazolam infusions) and demonstrated a rapid and robust improvement in PTSD symptoms. Median time to loss of response, however, occurred a few weeks following the course of infusions, making it imperative to investigate novel approaches aimed at preventing symptom relapse following ketamine treatment. The study team proposes a proof-of-concept, open-label pilot study to evaluate the efficacy of adding an evidence-based, brief and scalable trauma-focused psychotherapy, Written Exposure Therapy (WET), to a course of ketamine infusions in improving PTSD symptoms and maintaining symptom improvement, in participants with chronic PTSD. To accomplish this aim, the study team will enroll individuals who meet DSM-5 criteria for chronic PTSD. Eligible patients will receive a total of six ketamine infusions and will participate in WET (a total of five sessions). The primary outcome will be change in PTSD symptom severity from baseline to 12 weeks from the start of WET, assessed with the Clinician-Administered PTSD Scale for DSM-5. Additionally, all participants will be assessed weekly until 12 weeks following the start of WET. Thereafter, participants who remain improved will be assessed monthly for up to 24 weeks. The study team will also evaluate whether extinction learning ability -assessed with a computerized extinction learning task- predicts maintenance of ketamine response over time, and will explore potential sociodemographic and clinical predictors of treatment response. If demonstrated to have preliminary efficacy, this novel combined treatment may represent a promising intervention for individuals with chronic PTSD, deserving further study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 18-70 years of age;
2. Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document;
3. Participants must fulfill DSM-5 criteria for current civilian or combat-related PTSD, based on clinical assessment by a study psychiatrist and on the CAPS-5, and a past-month total CAPS5 score ≥ 30 at screening - this is done to ensure at least moderate severity and to safeguard against high placebo response rates;
4. Women must be using a medically accepted reliable means of contraception (if using an oral contraceptive medication, they must also be using a barrier contraceptive) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year);
5. Women of childbearing potential must have a negative pregnancy test at screening and prior to each intravenous infusion;
6. Men who are sexually active with women of childbearing potential must use a medically accepted reliable means of contraception and must agree not to donate sperm for a period of 90 days after receiving the last dose of ketamine;
7. Participants must be able to identify a family member, physician, or friend (i.e. someone who knows them well) who will participate in a Treatment Contract (and e.g. contact the study physician on their behalf in case manic symptoms or suicidal thoughts develop).

Exclusion Criteria:

1. Women who plan to become pregnant, are pregnant or are breast-feeding (because the medical risk of using ketamine during pregnancy and breast-feeding is unknown);
2. Serious, unstable medical illnesses such as hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, including gastro-esophageal reflux disease, obstructive sleep apnea, history of difficulty with airway management during previous anesthetics, ischemic heart disease and uncontrolled hypertension, and history of severe head injury;
3. Clinically significant abnormal findings of laboratory parameters, physical examination, or ECG;
4. Renal impairment, as reflected by a BUN >20 mg/dL, and/or creatinine clearance of >1.3 mg/dL;
5. Clinically significant uncorrected hypothyroidism or hyperthyroidism, as indicated by a TSH value 25% above or below the normal range;
6. A Body Mass Index (BMI) >40;
7. Hormonal treatment (e.g., estrogen) started in the 3 months prior to the first infusion day;
8. History of a neurodevelopmental disorder (e.g., autism, pervasive developmental disorder) ;
9. History of one or more seizures without a clear and resolved etiology;
10. Lifetime history of bipolar I or II disorder;
11. Presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia or schizoaffective disorder;
12. Drug or alcohol use disorder within the preceding 3 months
13. Previous recreational use of ketamine or PCP on more than one occasion, or any recreational use of ketamine or PCP within the last two years;
14. Previous non-response to clinical or research ketamine or esketamine administration;
15. Current diagnosis of bulimia nervosa or anorexia nervosa;
16. Patients judged clinically to be at serious and imminent suicidal or homicidal risk;
17. SBP >165 and DBP >95 at infusion days - higher BP allowed to account for stress or anxiety;
18. Concurrent treatment with opioid medication, or with long-acting or daytime short-acting benzodiazepines within two weeks of study start;
19. Current cognitive impairment, as defined by a score <23 on the Montreal Cognitive Assessment (MoCA);
20. Estimated IQ <80;
21. Currently receiving evidence-based psychotherapy for PTSD (e.g., prolonged exposure, cognitive processing therapy);

Note: Concurrent treatment with other psychotropic medications (including a short-acting benzodiazepine at bedtime only) will be permitted, but dose must be stabilized for at least three months before study start.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Feder, MD, Principal Investigator — Depression and Anxiety Center, Icahn School of Medicine at Mount Sinai; Oneysha Brown, BA, Study Director — Depression and Anxiety Center, Icahn School of Medicine at Mount Sinai
Locations (1):
- Depression and Anxiety Center, Icahn School of Medicine at Mount Sinai, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Upon receipt of request by PI, and after obtaining the necessary Data Transfer Agreement, PI will provide requested de-identified data via CSV file.

REFERENCES:
- [Derived] Feder A, Brown O, Rutter SB, Cahn L, Overbey JR, Seeley SH, Yu A, Bonanno PA, Fremont RA, Delgado AA, Jha MK, Costi S, Yehuda R, Schiller D, Pietrzak RH, Charney DS, Sloan DM, Murrough JW. Combining Ketamine Infusions and Written Exposure Therapy for Chronic PTSD: An Open-Label Trial. J Clin Psychiatry. 2025 Apr 2;86(2):24m15622. doi: 10.4088/JCP.24m15622. PMID 40215385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants signed consent and considered enrolled
Period: Screen
Arm/Group | Ketamine and Written Exposure Therapy
Started | 16
Completed | 14
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Failed to meet screening criteria | 1
Period: Study Treatment
Arm/Group | Ketamine and Written Exposure Therapy
Started | 14
Completed | 13
Not Completed | 1
Not completed — Exited by study team due to inappropriate behavior | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine and Written Exposure Therapy
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 1
Duration of PTSD [Mean (Standard Deviation); unit: years] | 18.1 (14)
Number of Participants taking Concomitant treatment with psychotropic medication [Count of Participants; unit: Participants] | 6
Clinician Administered PTSD Scale (CAPS-5) score [Mean (Standard Deviation); unit: units on a scale] — Past month, reported at screening visit (1-2 months prior to baseline visit)
  CAPS is a 30-item structured diagnostic interview designed to measure frequency and intensity of PTSD symptoms. The symptoms are scored in a 0-4 Likert-type scale, total score ranging from 0 to 80, higher score indicates more symptoms
  units on a scale | 40.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: CAPS-5
Description: Clinician Administered PTSD Scale for DSM-5 (CAPS-5), assessed at baseline (before the first infusion) and 12 weeks following the start of WET. The Clinician-Administered PTSD Scale (CAPS) is a 30-item structured diagnostic interview designed to measure frequency and intensity of PTSD symptoms. The symptoms are scored in a 0-4 Likert-type scale, total score ranging from 0 to 80, higher score indicates more symptoms
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine and Written Exposure Therapy
Number analyzed (Participants) | 13
score on a scale
  Baseline, the morning of first ketamine infusion | 41.6 (6.2)
  Week 12 | 20.8 (14.8)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Ketamine and Written Exposure Therapy
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketamine and Written Exposure Therapy (N=13)
Nausea/vomiting (Gastrointestinal disorders) | 2
Increased Perspiration (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 5
Blurred Vision (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 5
Frequent Urination (Renal and urinary disorders) | 2
Difficulty Sleeping (General disorders) | 2
Menstrual Irregularity (Reproductive system and breast disorders) | 2
Fatigue (General disorders) | 11
Decreased energy (General disorders) | 1
Anxiety (General disorders) | 1
Other (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04889664/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04889664/ICF_001.pdf